CLINICAL TRIAL: NCT06370026
Title: KSD-101 Therapy for Standard Treatment Failed EBV-associated Nasopharyngeal Carcinoma: an Exploratory Clinical Trial
Brief Title: KSD-101 Therapy for Standard Treatment Failed EBV-associated NPC: an Exploratory Clinical Trial
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Kousai Bio Co., Ltd. (Other)
Responsible Party: Principal Investigator, Fei Han, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSD-101-CR004
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: EBV; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KSD-101 (Experimental): Biological: Dendritic Cell Vaccine.Autologous monocyte-derived DCs pulsed with EBV antigen.
  Interventions: Biological: KSD-101

INTERVENTIONS:
Biological: KSD-101 — Patients will receive approximately 5x10^6 DC vaccine via subcutaneous injections bi-weekly,total 3-5 times.

SUMMARY:
The main purpse of this study is to evaluate the safety of KSD-101 in patients with EBV-associated Nasopharyngeal Carcinoma,to evaluate the initial clinical outcomes and evaluate the immune response to KSD-101 for the treatment in Patients with EBV-associated Nasopharyngeal Carcinoma.

DETAILED DESCRIPTION:
This is a single-center, single-arm, open, multiple-dose clinical study evaluating the safety, preliminary efficacy, and immune response of KSD-101 for the treatment of patients with EBV-associated nasopharyngeal carcinoma.

Approximately 120 mL of PBMCs is collected from subjects. The collected PBMCs are transported to the manufacturing facility for the preparation of KSD-101. Subjects return to the study site for subsequent visits at investigator-notified times.

1. KSD-101 route of administration: subcutaneous injection.
2. KSD-101 treatment dose: 5.0 × 10^6 cells/dose.
3. KSD-101 treatment frequency: once every 2 weeks for a total of 3-5 times. The 4th and 5th times are booster treatments, which need to be decided by the investigator according to the condition of the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their legal guardian voluntarily participate and sign an informed consent form.
2. Female or emale patients aged 18-70 years (inclusive of the cut-off value) on the date of signing the informed consent.
3. Nasopharyngeal carcinoma confirmed by pathological tissue examination and EBER-positive in tumor tissue by in situ hybridization (ISH or FISH).
4. Nasopharyngeal carcinoma that has failed 3rd or more line treatment and has localized recurrence or localized recurrence with systemic metastasis or primary metastatic nasopharyngeal carcinoma that is not suitable for localized or radical treatment.
5. At least one measurable lesion according to RECIST v1.1 criteria.
6. An Eastern Cooperative Oncology Group (ECOG) score of 0 to 1.
7. Have criteria for single or venous blood collection and have no other contraindications to cell collection.
8. Patients' laboratory findings are compatible:

   * Blood routine: neutrophils ≥ 1.5×10^9/L, hemoglobin ≥ 90g/L, platelets ≥ 100×10^9/L.
   * Liver function: ALT, AST ≤ 3 × ULN and total bilirubin ≤ 1.5 × ULN.
   * Renal function: creatinine ≤ 1.5 × ULN.
   * Cardiac function: left ventricular ejection fraction (LVEF) ≥ 40%.
   * Coagulation function: fibrinogen ≥ 1.0g/L, activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, prothrombin time (PT) ≤ 1.5 × ULN.
9. Patients' corresponding lymph node region can accommodate subcutaneous injections.
10. Expected survival ≥ 3 months.

Exclusion Criteria:

1. Patients receiving any anti-tumor therapy such as chemotherapy, radiotherapy, immunosuppressive therapy, etc. within 4 weeks prior to mono-collection.
2. Women who are pregnant (positive urine/blood pregnancy test), breastfeeding, or men or women who are planning to conceive within the last 1 year.
3. Active hepatitis B (HbsAg or HbcAb positive and HBV DNA ≥100 IU/mL), active hepatitis C (HCV antibody positive and peripheral blood HCV RNA positive); human immunodeficiency virus (HIV) antibody positive; syphilis test positive.
4. Patients with central nervous system pathology (e.g., cerebral edema, need for hormonal intervention, or progression of brain metastases).
5. Patients with uncontrollable infectious disease within 4 weeks prior to enrollment, or with active tuberculosis or on anti-tuberculosis therapy. (< CTCAE grade 2 genitourinary infections and upper respiratory tract infections, except EBV infections).
6. Patients have a serious underlying disease (cardiovascular disease, respiratory disease, renal insufficiency, coagulation abnormality, autoimmune disease or immunodeficiency disease, etc.).
7. Other active malignant tumors within the past 3 years, unless they are curable tumors and have been significantly cured, such as basal or squamous cell carcinoma, carcinoma in situ of the uterine cervix or breast.
8. Subjects who have undergone major surgery or severe trauma within 4 weeks prior to enrollment or are expected to require major surgical intervention (i.e., surgery requiring the assistance of endotracheal anesthesia) during the study period.
9. Patients have received a prophylactic live or live attenuated vaccine within 4 weeks prior to screening.
10. Patients have participated in another clinical study within 4 weeks prior to screening.
11. Patients with a prior history of severe drug allergy, or penicillin allergy.
12. Patients have substance abuse/addiction.
13. Patients have other conditions that, in the judgment of the investigator, make enrollment inappropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence Adverse events (Safety endpoint) | 1 year after DC Vaccines injection
  Adverse events will be graded according to the NCI-CTCAE 5.0 grading criteria throughout the study period, except for injection site (localized) adverse events, which will be graded with reference to the Guidelines for Grading Criteria for Adverse Events in Clinical Trials of Vaccines for Prophylaxis.

SECONDARY OUTCOMES:
EBV-DNA load | 1 year after DC Vaccines injection
  changes in EBV-DNA load were assessed during the study
Objective response rate (ORR) | 1 year after DC Vaccines injection
  The percentage of participants who achieved PR or better response
Disease control rate (DCR) | 1 year after DC Vaccines injection
  The percentage of participants who achieved SD or better response
Duration of response (DOR) | 1 year after DC Vaccines injection
  DOR will be calculated among responders (with a PR or better response) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease
Progression-free survival (PFS) | 1 year after DC Vaccines injection
  The time from the start of CAR-GPRC5D treatment for the participants to the first time of disease progression or death for any reason
Overall survival (OS) | 1 year after DC Vaccines injection
  OS is measured from the date of the initial injection of DC Vaccines to the date of the participant's death
Levels of EBV-specific CD8+ T cells | 1 year after DC Vaccines injection
  EBV-specific CD8+ T cells in peripheral blood will be assessed to monitor changes
Levels of B cells | 1 year after DC Vaccines injection
  B cells in peripheral blood will be assessed to monitor changes
Levels of NK cells | 1 year after DC Vaccines injection
  NK cells in peripheral blood will be assessed to monitor changes
According to EORTC QLQ-C30 | Up to 1 year
  Changes of Quality of life, according to EORTC QLQ-C30
According to EQ-5D-5L | Up to 1 year
  Changes of Quality of life, according to EQ-5D-5L
According to EORTC QLQ-H&N35 | Up to 1 year
  Changes of Quality of life, according to EORTC QLQ-H&N35
According to ECOG fitness status | Up to 1 year
  Changes of Quality of life, according to ECOG fitness status

CONTACTS AND LOCATIONS:
Overall Officials: Fei Han, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No